CLINICAL TRIAL: NCT06992596
Title: UAE-PRIME: A Feasibility Study of a Precise Robotically Implanted Brain-Computer Interface for the Control of External Devices
Acronym: UAE-PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralink Corp (Industry)
Collaborators: Cleveland Clinic Abu Dhabi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: N1-FS-001; ADHRTC-2025-65 (Other: Department of Health)
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Tetraplegia/Tetraparesis; Quadriplegia; Quadriplegia/Tetraplegia; Cervical Spinal Cord Injury; Amyotrophic Lateral Sclerosis (ALS); Spinal Cord Injury (Quadraplegia); Spinal Cord Injury; Motor Neuron Disease; Brain Stem Stroke
Keywords: brain computer interface; Neuralink N1 Implant; Neuralink; Robot; tetraparesis; tetraplegia; quadriplegia; ALS; spinal cord injury; Amyotrophic lateral sclerosis; chip; brain chip; External device control; Wireless implant; Neuroprosthetics; SCI; paralysis; motor neuron disease
MeSH Terms: conditions — Quadriplegia; Amyotrophic Lateral Sclerosis; Spinal Cord Injuries; Motor Neuron Disease; Brain Stem Infarctions; Paralysis

STUDY DESIGN:
Intervention Model Description: The study is a prospective, longitudinal, open-label, single-arm feasibility study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UAE-PRIME: Precise Robotically Implanted Brain-Computer Interface (Other): Open label
  Interventions: Device: N1 Implant; Device: R1 Robot

INTERVENTIONS:
Device: N1 Implant — The N1 Implant is a type of implantable brain-computer interface.
Device: R1 Robot — The R1 Robot is a robotic electrode thread inserter that implants the N1 Implant.

SUMMARY:
The UAE-PRIME Study is a feasibility study designed to assess the initial clinical safety and functionality of the Neuralink N1 Implant and R1 Robot. This study involves participants who have tetraparesis, tetraplegia, or a diagnosis that may lead to these conditions.

The N1 Implant is a wireless, rechargeable device mounted on the skull, connected to electrode threads that are inserted into the brain by the R1 Robot, which is a robotic device specifically designed for this procedure.

ELIGIBILITY:
Inclusion Criteria:

* (a) A diagnosis of a spinal cord injury (>12 months), stroke (>12 months), or other neurological condition causing the participant to experience bilateral upper limb motor impairment, with no expectation of recovery.

OR (b) A diagnosis of Amyotrophic Lateral Sclerosis (ALS) or other progressive neurological condition where the natural history of the disease is well understood and where there is tetraparesis and the expectation, in the view of the participant's treating neurologist, that the disease will progress such that the participant will meet criteria 1a within 1 year of recruitment.

* Life expectancy ≥ 12 months.
* Ability to communicate verbally or with the use of a computer or communication aid, and working proficiency in English.
* Presence of a stable caregiver

Exclusion Criteria:

* Moderate to high risk for serious perioperative adverse events
* Morbid obesity (Body Mass Index > 40)
* History of poorly controlled seizures or epilepsy
* History of poorly controlled diabetes
* Requires magnetic resonance imaging (MRI) for any ongoing medical conditions
* Acquired or hereditary immunosuppression
* Smoking tobacco or use of other tobacco products > once per month within the last year.
* Psychiatric or psychological disorder
* Pre-existing damage to the cortical region of interest (as determined by MRI)
* Any condition which, in the opinion of the Investigator, would compromise your ability to safely participate in the study or undergo the implantation procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
The Rate of Device-Related Adverse Events (AE) | 12 months post-implant
The Rate of Procedure-Related Adverse Events (AE) | 12 months post-implant

SECONDARY OUTCOMES:
The Rate of Device-Related Adverse Events (AE) | Up to 36 months post-implant
The Rate of Procedure-Related Adverse Events (AE) | Up to 36 months post-implant
Change in Montreal Cognitive Assessment (MoCA) score during the Primary Study | From baseline to 30-days, 3-, 6-, 9-, and 12-months post-implantation
  The Montreal Cognitive Assessment (MoCA) is a 30-point scale assessing cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive performance. Outcome will be reported as change from baseline at each follow-up visit.
Change in Montreal Cognitive Assessment (MoCA) score during the Long-term Follow-up Phase | From baseline to 36-months post-implantation
  The Montreal Cognitive Assessment (MoCA) is a 30-point scale assessing cognitive function. Scores range from 0 to 30, with higher scores indicating better cognitive performance. Outcome will be reported as change from baseline at each follow-up visit.
Change in Patient Health Questionnaire-9 (PHQ-9) score during the Primary Study | From baseline to 30-days, 3-, 6-, 9-, and 12-months post-implantation
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale used to assess depression severity. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. Outcome will be reported as change from baseline at each follow-up visit.
Change in Patient Health Questionnaire-9 (PHQ-9) score during the Long-term Follow-up Phase | From baseline to 36-months post-implantation
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item scale used to assess depression severity. Scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. Outcome will be reported as change from baseline at each follow-up visit.
Change in Generalized Anxiety Disorder-7 (GAD-7) score during the Primary Study | From baseline to 30-days, 3-, 6-, 9-, and 12-months post-implantation
  The Generalized Anxiety Disorder 7-item (GAD-7) scale assesses anxiety severity. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. Outcome will be reported as change from baseline at each follow-up visit.
Change in Generalized Anxiety Disorder-7 (GAD-7) score during the Long-term Follow-up Phase | From baseline to 36-months post-implantation
  The Generalized Anxiety Disorder 7-item (GAD-7) scale assesses anxiety severity. Scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. Outcome will be reported as change from baseline at each follow-up visit.
Change in neurological function as assessed by standardized physician neurological exam during the Primary Study | From baseline to 30-days, 3-, 6-, 9-, and 12-months post-implantation
  Neurological function will be assessed by a study physician using a standardized neurological exam covering motor strength, reflexes, coordination, cranial nerve function, and sensory status.
Change in neurological function as assessed by standardized physician neurological exam during the Long-term Follow-up Phase | From baseline to 36-months post-implantation
  Neurological function will be assessed by a study physician using a standardized neurological exam covering motor strength, reflexes, coordination, cranial nerve function, and sensory status.

CONTACTS AND LOCATIONS:
Overall Officials: Florian Roser, MD, Principal Investigator — Cleveland Clinic Abu Dhabi
Locations (1):
- Cleveland Clinic Abu Dhabi (CCAD), Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuralink's Patient Registry — https://neuralink.com/patient-registry/
- See also: Neuralink Website — https://neuralink.com/